CLINICAL TRIAL: NCT01401010
Title: Pharmacokinetic/Pharmacodynamic Study of Doripenem in Febrile Neutropenic Patients With Possible Bacterial Infection
Brief Title: Pharmacokinetic/Pharmacodynamic Study of Doripenem in Febrile Neutropenic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gary E. Stein, Pharm.D. (Other)
Responsible Party: Sponsor-Investigator, Gary E. Stein, Pharm.D., Professor of Medicine and Pharmacology, Michigan State University
Organization: Michigan State University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DORIBAC4006a
Record Dates: First submitted 2011-07-14; First posted 2011-07-25 (Estimated); Results first posted 2012-06-05 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Febrile Neutropenia
Keywords: neutropenia; doripenem
MeSH Terms: conditions — Febrile Neutropenia; Neutropenia | interventions — Doripenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doripenem 500 mg (Active Comparator): pharmacokinetics/pharmacodynamics
  Interventions: Drug: Doripenem
- Doripenem 1000 mg (Active Comparator): pharmacokinetics/pharmacodynamics
  Interventions: Drug: doripenem

INTERVENTIONS:
Drug: Doripenem — 500 mg every 8 hours
  Other Names: Doribac
  Arms: Doripenem 500 mg
Drug: doripenem — 1000 mg every 8 hours
  Other Names: Doribac
  Arms: Doripenem 1000 mg

SUMMARY:
Primary: To determine the serum pharmacokinetics (PK) of doripenem in febrile neutropenic patients.

Secondary: Monte Carlo Simulations Tested Against Various Gram-negative Isolates and Reported as Probability of Target Attainment (40% Time (fT)> minimum inhibitory concentration (MIC))

DETAILED DESCRIPTION:
Background: Doripenem is a group 2 carbapenem with enhanced in vitro activity against Gram-negative bacteria including Pseudomonas aeruginosa. Currently, there is a paucity of pharmacokinetic/pharmacodynamic data on doripenem in patients with febrile neutropenia.

Objectives: To conduct a pharmacokinetic and safety evaluation of two doses of doripenem in febrile neutropenic patients and provide probability estimates of attaining effective drug exposure against common Gram-negative pathogens.

Methods: We obtained multiple blood samples from 12 adult patients with febrile neutropenia who were receiving either 500 mg or 1000 mg of doripenem IV over 4-hours every 8 hours. Following at least 2 doses, serum concentrations were measured in each subject at 1, 4, 6 and 8 hours after initiation of a dose by a validated HPLC assay. The derived pharmacokinetic (PK) parameters from these serum levels were utilized to perform a 5000 patient Monte Carlo simulation against bacteria with minimal inhibitory concentrations (MICs) of 0.008 to 64 mg/L to determine probability estimates of time of free drug concentration > MIC (fT>MIC).

Results: The mean PK parameters in these patients were a volume of distribution (Vd) of 43.9L, an elimination rate constant (k) of 0.37 hr -1, a total clearance (Cl) of 14.4 L/h, and an area under the concentration-time curve (AUC) of 57.6 mg∙h/L. An optimal probability of target attainment (40% fT>MIC) of 90% was obtained against bacteria with MICs ≤ 2.0 and ≤ 4.0 mg/L with 500 mg and 1000 mg doses, respectively. Adverse events associated with doripenem were not observed in these patients.

Conclusions: The findings from this analysis of doripenem suggest that higher doses as well as prolonged infusions may be necessary to optimally treat selected Gram-negative bacteria (eg. Pseudomonas aeruginosa) in patients with febrile neutropenia

ELIGIBILITY:
Inclusion Criteria:

* adult neutropenic (< 500 cells) patients who are febrile

Exclusion Criteria:

* Patients with Creatinine Clearance < 30 ml/min or allergy to carbapenems will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Stein, PharmD, Principal Investigator — Michigan State University
Locations (1):
- Sparrow Hospital, Lansing, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were inpatients (Sparrow Hospital) with febrile neutropenia who were treated with doripenem; referral base was infectious disease consultations. The first patient was enrolled 6-15-2010 and the last 8-21-2011.
Period: Overall Study
Arm/Group | Doripenem 500 mg | Doripenem 1000 mg
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Could not interpret assay results | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doripenem 500 mg | Doripenem 1000 mg | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (17) | 49 (18) | 49 (17.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean (SD) Doripenem Pharmacokinetic Volume of Distribution Parameter in Febrile Neutropenic Patients
Description: To determine the serum pharmacokinetic volume of distribution of doripenem in febrile neutropenic patients with pneumonia. We obtained blood at 1, 4, 6, 8 hours after at least two doses of doripenem and measured these levels (mg/L)by HPLC assay.
Time Frame: 1, 4, 6, 8 hours after at least two doses of drug
Population: Each subject received drug and had serum samples drawn at 1, 4, 6, 8 hours after dosing.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Doripenem 500 mg: Mean (SD) Doripenem Pharmacokinetic (PK) Parameters in Febrile Neutropenic Patients Who Received 500mg Dosing
- Doripenem 1000 mg: Mean (SD) Doripenem Pharmacokinetic (PK) Parameters in Febrile Neutropenic Patients Who Received 1000 mg Dosing
- Combined Results for Both 500 and 1000 mg: Mean (SD) Doripenem Pharmacokinetic (PK) Parameters in Febrile Neutropenic Patients Combined Results
Arm/Group | Doripenem 500 mg | Doripenem 1000 mg | Combined Results for Both 500 and 1000 mg
Number analyzed (Participants) | 5 | 6 | 11
Liters | 36.7 (15.9) | 49.9 (18.1) | 43.9 (17.7)

2. Secondary Outcome: Monte Carlo Simulations Tested Against Various Gram-negative Isolates and Reported as Probability of Target Attainment (40% Time (fT) > Minimum Inhibitory Concentrations (MIC))
Description: Following determination of pharmacokinetic (PK) parameters from patients with febrile neutropenia, Monte Carlo simulations were then conducted to determine time of serum concentrations above the MIC (40% of the time) against Gram-negative isolates.
  These Gram-negative isolates had a range of minimum inhibitory concentrations (MIC) to Doripenem.
Time Frame: 1, 4, 6, 8 hours after an infusion of doripenem to determine the PK parameters
Population: Each subject received drug and had serum samples drawn at 1, 4, 6, 8 hours after dosing.
Measure: Number; unit: probability of target attainment
Groups:
- 500 mg Doripenem 1 Hour Infusion; 500 mg Doripenem 4 Hour Infusion; 1000 mg Doripenem 1 Hour Infusion; 1000 mg Doripenem 4 Hour Infusion: Probability of target attainment (40%fT>MIC) against Gram-negative pathogens using Monte Carlo simulations
Arm/Group | 500 mg Doripenem 1 Hour Infusion | 500 mg Doripenem 4 Hour Infusion | 1000 mg Doripenem 1 Hour Infusion | 1000 mg Doripenem 4 Hour Infusion
Number analyzed (Participants) | 5 | 5 | 6 | 6
probability of target attainment
  E. coli MIC: 0.06 mg/L | 1 | 1 | 1 | 1
  K. pneumoniae MIC: 0.12 mg/L | 0.99 | 1 | 1 | 1
  P. mirabilis MIC: 0.50 mg/L | 0.99 | 1 | 0.99 | 1
  E. cloacae MIC: 0.25 mg/L | 0.99 | 1 | 0.99 | 1
  S. marcescens MIC: 0.25 mg/L | 0.99 | 1 | 0.99 | 0.99
  P. aeruginosa MIC: 4 mg/L | 0.55 | 0.63 | 0.87 | 0.94

3. Primary Outcome: Mean (SD) Doripenem Pharmacokinetic (PK) Elimination Rate Constant Parameter in Febrile Neutropenic Patients
Description: To determine the serum pharmacokinetic elimination rate constant of doripenem in febrile neutropenic patients with pneumonia. We obtained blood at 1, 4, 6, 8 hours after at least two doses of doripenem and measured these levels (mg/L)by HPLC assay.
Time Frame: 1, 4, 6, 8 hours after at least two doses of drug
Population: Each subject received drug and had serum samples drawn at 1, 4, 6, 8 hours after dosing.
Measure: Mean (Standard Deviation); unit: hour^-1
Arm/Group | Doripenem 500 mg | Doripenem 1000 mg | Combined Results for Both 500 and 1000 mg
Number analyzed (Participants) | 5 | 6 | 11
hour^-1 | 0.36 (0.14) | 0.38 (0.20) | 0.37 (0.17)

4. Primary Outcome: Mean (SD) Doripenem Pharmacokinetic (PK) Half Life Parameter in Febrile Neutropenic Patients
Description: To determine the serum pharmacokinetic half life of doripenem in febrile neutropenic patients with pneumonia. We obtained blood at 1, 4, 6, 8 hours after at least two doses of doripenem and measured these levels (mg/L)by HPLC assay.
Time Frame: 1, 4, 6, 8 hours after at least two doses of drug
Population: Each subject received drug and had serum samples drawn at 1, 4, 6, 8 hours after dosing.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Doripenem 500 mg | Doripenem 1000 mg | Combined Results for Both 500 and 1000 mg
Number analyzed (Participants) | 5 | 6 | 11
hours | 2.2 (0.84) | 2.4 (1.3) | 2.3 (1.1)

5. Primary Outcome: Mean (SD) Doripenem Pharmacokinetic (PK) Clearance of Drug Parameter in Febrile Neutropenic Patients
Description: To determine the serum pharmacokinetic clearance of drug of doripenem in febrile neutropenic patients with pneumonia. We obtained blood at 1, 4, 6, 8 hours after at least two doses of doripenem and measured these levels (mg/L)by HPLC assay.
Time Frame: 1, 4, 6, 8 hours after at least two doses of drug
Population: Each subject received drug and had serum samples drawn at 1, 4, 6, 8 hours after dosing.
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | Doripenem 500 mg | Doripenem 1000 mg | Combined Results for Both 500 and 1000 mg
Number analyzed (Participants) | 5 | 6 | 11
Liters/hour | 11.9 (2.2) | 16.6 (6.8) | 14.4 (5.6)

6. Primary Outcome: Mean (SD) Doripenem Pharmacokinetic (PK) Area Under Serum Curve (mg*h/L) Parameter in Febrile Neutropenic Patients
Description: To determine the serum pharmacokinetic area under serum curve of doripenem in febrile neutropenic patients with pneumonia. We obtained blood at 1, 4, 6, 8 hours after at least two doses of doripenem and measured these levels (mg/L)by HPLC assay.
Time Frame: 1, 4, 6, 8 hours after at least two doses of drug
Population: Each subject received drug and had serum samples drawn at 1, 4, 6, 8 hours after dosing.
Measure: Mean (Standard Deviation); unit: milligrams * hour/liters
Arm/Group | Doripenem 500 mg | Doripenem 1000 mg | Combined Results for Both 500 and 1000 mg
Number analyzed (Participants) | 5 | 6 | 11
milligrams * hour/liters | 47.1 (13.2) | 66.4 (33.1) | 57.6 (26.8)

ADVERSE EVENTS:
Arm/Group | Doripenem 500 mg | Doripenem 1000 mg
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No